CLINICAL TRIAL: NCT03912636
Title: Rumination Syndrome: Role of Vagal Tone and Effect of Respiratory Manoeuvres on Severity and Frequency of Rumination
Brief Title: Role of Vagal Tone in Rumination Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19/ss/0054
Record Dates: First submitted 2019-03-26; First posted 2019-04-11 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Rumination
Keywords: cardiac vagal tone; deep breathing; diaphragmatic breathing; vagal nerve; vagal tone; cognitive behavioral therapy; visceral hypersensitivity
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: In study 1 for the pathophysiology of rumination syndrome, the investigators will recruit 10 healthy volunteers and 10 patients. In study 2 for the treatment, the investigators will recruit 10 patients and perform the cross-over test, in which the patients will perform 2 breathing exercises and the investigators will compare the effects.
Masking Description: When the investigators analyze the data, the investigator will be blinded to the conditions of the participants and the types of breathing exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Diaphragmatic breathing in healthy volunteers in study1 (Active Comparator): Healthy volunteers will perform diaphragmatic breathing, and the investigators will investigate changes of cardiac vagal tone.
  Interventions: Behavioral: Diaphragmatic breathing
- Diaphragmatic breathing in rumination patients in study1 (Active Comparator): Rumination patients will perform diaphragmatic breathing, and the investigators will investigate changes of cardiac vagal tone.
  Interventions: Behavioral: Diaphragmatic breathing
- Deep slow breathing in healthy volunteers in study1 (Active Comparator): Healthy volunteers will perform deep slow breathing, and the investigators will investigate changes of cardiac vagal tone.
  Interventions: Behavioral: Deep Slow Breathing
- Deep slow breathing in rumination patients in study1 (Active Comparator): Rumination patients will perform deep slow breathing, and the investigators will investigate changes of cardiac vagal tone.
  Interventions: Behavioral: Deep Slow Breathing
- Normal breathing in healthy volunteers in study1 (Placebo Comparator): healthy volunteers will perform normal breathing, and the investigators will investigate changes of cardiac vagal tone.
  Interventions: Behavioral: Normal breathing
- Normal breathing in rumination patients in study1 (Placebo Comparator): rumination patients will perform normal breathing, and the investigators will investigate changes of cardiac vagal tone.
  Interventions: Behavioral: Normal breathing
- Diaphragmatic breathing in study 2; cross over test (Active Comparator): Rumination patients will perform diaphragmatic breathing in randomized cross-over test. The investigators will compare the effects on rumination.
  Interventions: Behavioral: Diaphragmatic breathing
- Deep slow breathing in study 2; cross over test (Active Comparator): Rumination patients will perform diaphragmatic breathing in randomized cross-over test. The investigators will compare the effects on rumination.
  Interventions: Behavioral: Deep Slow Breathing

INTERVENTIONS:
Behavioral: Diaphragmatic breathing — Subjects will perform Diaphragmatic breathing after the test meal.
  Arms: Diaphragmatic breathing in healthy volunteers in study1; Diaphragmatic breathing in rumination patients in study1; Diaphragmatic breathing in study 2; cross over test
Behavioral: Deep Slow Breathing — Subjects will perform Deep Slow Breathing after the test meal.
  Arms: Deep slow breathing in healthy volunteers in study1; Deep slow breathing in rumination patients in study1; Deep slow breathing in study 2; cross over test
Behavioral: Normal breathing — Subjects will perform Normal Breathing (as a control) after the test meal as a control.
  Arms: Normal breathing in healthy volunteers in study1; Normal breathing in rumination patients in study1

SUMMARY:
Rumination syndrome is a condition in which people repeatedly and unintentionally regurgitate undigested or partially digested food from the stomach, rechew it, and then either re-swallow it or spit it out. The mechanism of the disease is not well understood. The investigators believe that discomfort in the stomach during and immediately after meals may be an important factor for this disease. The reason for such discomfort can be due to an alteration of nervous regulation of the stomach. The investigators can study the nervous regulation that affects the stomach and other parts of the body by analysing in detail an electrocardiogram that is performed continuously for several hours. From this analysis, The investigators can study a parameter called cardiac vagal tone (CVT).

Diaphragmatic breathing (DiaB) is a respiratory exercise, in which people mainly move their abdomen to breath. DiaB is a common treatment for rumination syndrome. Patients doing DiaB can reduce the number of rumination episodes. The mechanism by which DiaB improves rumination is unknown. There is another type of breathing called slow deep breathing (SlowDB), in which people mainly breathe with their chest. SlowDB is used as a therapy for increased pain in the food pipe (oesophagus) and it might also be effective on rumination syndrome. The investigators believe that both DiaB and SlowDB can improve rumination, by modifying the nervous control of the stomach (that the investigators can monitor by measuring continuously cardiac vagal tone (CVT)). The aims of the study are to investigate the association between gastric discomfort during a meal, CVT variations (measured with the electrocardiogram during the meal) and the severity of rumination episodes. The investigators will also study how DiaB and SlowDB can modify this variable during the test. In a second step, The investigators will assess the clinical effect of respiratory exercises (DiaB and SlowDB) on the severity and frequency of regurgitations in patients diagnosed with rumination syndrome.

Method This research consists of two separate studies.

1. Study1 (to investigate the mechanism of rumination syndrome) 10 healthy volunteers and 10 rumination patients will join Study1 on 3 separate days. On each visit, the investigators will place electrocardiogram sensors and a belt that can measure the thorax or abdominal movement. All subjects will get instructions to perform SlowDB or DiaB, answer some questionnaires, eat the test meal, perform normal breathing/DiaB/SlowDB for 15 minutes, and stay quietly on the chair for 3 hours.
2. Study 2 (to assess the effect of DiaB and SlowDB on rumination syndrome) 10 patients with rumination syndrome will join Study 2. On the first visit, subjects will have the test meal, answer the symptom questionnaire 1 hour after the meal, and learn how to perform either DiaB or SlowDB. After the first visit, subjects perform DiaB or SlowDB during 15 minutes after every meal for 4 weeks. On the second visit, subjects will have the test meal, answer the symptom questionnaire 1 hour after the meal, and learn how to perform the other respiratory exercise. After a 2-week break, subjects will perform the other respiratory exercise for the next 4 weeks. On the last visit, subjects will have the test meal and answer the symptom questionnaire 1 hour after the meal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers (HVs)

   * 18-65 years old
   * No history of any gastrointestinal (GI) symptoms in the 3 months prior to the study.
   * No medications 3 months prior to the study
2. Rumination patients

   * 18-65 years old
   * Fulfilling ROME IV clinical criteria for rumination
   * Confirmed rumination syndrome by High Resolution Impedance Monometry within 12 months prior to the study
   * No history of performing DiaB as a therapy for rumination syndrome.
   * No medications which may affect vagal tone, the number of rumination episodes and GI motility 3 months prior to the study. (i.e. opioids, Baclofen , anticholinergics drugs, prokinetics, beta-blockers)

Exclusion Criteria:

* Pregnant or lactating women
* History of GI surgeries apart from appendectomy
* Alcohol or substance abuse, mental health illness
* Inability to obtain informed consent
* Non-fluent English speakers
* Participants with food intolerances or allergies that would not be able to take in the test meal (McDonalds Big Mac meal)
* Major comorbidities such as significant cardiac/pulmonary disease, cancer, life-threatening conditions or other life-limiting conditions
* Evidence of relevant organic diseases. (in endoscopy, CT.)
* Evidence of major esophageal motility disorders (Chicago classification ver3.0) (21)
* Known allergy to ECG electrodes or latex
* History of diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of changes in cardiac vagal tone (CVT) calculated from R-R intervals in electrocardiogram between healthy volunteers and rumination patients in Study 1 | from baseline to 3-hour postprandial period.
  CVT is calculated from R-R intervals in electrocardiogram and measured on a validated linear vagal scale, where 0 represents full atropinisation. The investigators will continuously measure CVT during the 15-min baseline period, 30-min meal period, 15-min intervention period, and 3-h postprandial period.
Comparison of changes in Meal-induced discomfort scores between healthy volunteers and rumination patients in Study 1 | baseline, every 5 minutes during the 30-min meal period, every 30 minutes during the 3-hour postprandial period
  This score consists of 3 visual analog scales (VAS) of the level of nausea, fullness and epigastric discomfort. Each scale is graded from 0 to 5, where score 0 represents no perception and score 5 represents an extremely uncomfortable sensation. A Total score can vary between 0 and 15.
Comparison of changes in the number of rumination episodes between Diaphragmatic breathing group and Deep slow breathing group in Study 2 | from baseline to after the 4-week intervention period
  Subjects will count the number of rumination episodes during 1-hour postprandial period in the laboratory.

SECONDARY OUTCOMES:
Comparison of changes in cardiac vagal tone (CVT) calculated from R-R intervals in electrocardiogram among 3 respiratory exercises in Study 1 | from baseline to 3-hour postprandial period.
  CVT is calculated from R-R intervals in electrocardiogram and measured on a validated linear vagal scale, where 0 represents full atropinisation. The investigators will continuously measure CVT during the 15-min baseline period, 30-min meal period, 15-min intervention period, and 3-h postprandial period.
Comparison of the number of rumination episodes among 3 respiratory exercises in rumination patients in Study 1 | Baseline, meal period, 15-min intervention period, and first 1-hour postprandial period
  The subjects will count the number of rumination episodes the 15-min baseline period, 30-min meal period, 15-min intervention period, and the first 1-hour postprandial period.
Comparison of Treatment Evaluation scores in 2 groups in Study 2 | Baseline and every week during the 4-week intervention period
  The subjects will rate the perception of their complaints compared to the pre-treatment period from -3 to +3: -3 totally unbearable, -2 much worse, -1 slightly worse, 0 no change, +1 slightly better, +2 much better, and +3 totally resolved).
Comparison of changes in Meal-induced discomfort scores among 3 respiratory exercises in Study 1 | baseline, every 5 minutes during the 30-min meal period, every 30 minutes during the 3-hour postprandial period
  This score consists of 3 visual analog scales (VAS) of the level of nausea, fullness and epigastric discomfort. Each scale is graded from 0 to 5, where score 0 represents no perception and score 5 represents an extremely uncomfortable sensation. Total scores can vary between 0 and 15.

CONTACTS AND LOCATIONS:
Overall Officials: Mays Jawad, Study Chair — Joint Research Management Office, Queen Mary, University of London
Locations (1):
- Wingate Institue, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The investigators will not share the data with other researchers outside of our team.